CLINICAL TRIAL: NCT03443479
Title: Retrospective Cohort Study of Patients With Type II (Hypercapnic) Respiratory Failure Treated With High-flow Oxygen Therapy Versus Non-invasive Ventilation With BiPAP
Brief Title: Comparison of High-flow Oxygen vs. BiPAP in Type II (Hypercapnic) Respiratory Failure
Status: Completed | Type: Observational
Sponsor: Hôpital de Verdun (Other)
Responsible Party: Sponsor
Other Study IDs: OF1
Record Dates: First submitted 2018-02-15; First posted 2018-02-23 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Respiratory Failure; Respiratory Insufficiency; Respiratory Tract Diseases; COPD; COPD Exacerbation; Pneumonia; Chronic Obstructive Pulmonary Disease
Keywords: Non invasive ventilation; BiPAP; High-Flow Oxygen Therapy; High-Flow Nasal Cannula; COPD; Hypercapnia; Hypercapnic Respiratory failure; Chronic obstructive Pulmonary Disease
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Tract Diseases; Pulmonary Disease, Chronic Obstructive; Pneumonia; Hypercapnia | interventions — Noninvasive Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients with type II ARF: All patients with type II respiratory failure that were deemed by the treating physician to require ventilatory support either with non-invasive ventilation (NIV) or High-Flow Nasal Cannula (HFNC).
  Interventions: Device: Non-Invasive Ventilation; Device: High-Flow Nasal Cannula

INTERVENTIONS:
Device: Non-Invasive Ventilation — Treatment with Non-Invasive Ventilation by BiPAP. Different BiPAP models are in use. Ventilation parameters set at the discretion of the treating physician.
  Other Names: BiPAP
Device: High-Flow Nasal Cannula — Treatment with a High-Flow Nasal Cannula. The Optiflow device by Fisher&Paykel used in all cases. Flow and fraction of inspired oxygen (FiO2) parameters at the discretion of the treating physician.
  Other Names: HFNC

SUMMARY:
A retrospective cohort study of all patients treated for type II (hypercapnic) respiratory failure with either High-Flow Oxygen Therapy or Non-Invasive Ventilation in a general adult hospital.

DETAILED DESCRIPTION:
We will compare various clinically relevant outcomes in patients treated for type II (hypercapnic) acute respiratory failure (ARF) with either High-Flow Nasal Cannula (HFNC) or Non-Invasive Ventilation (NIV) in a general adult hospital.

All patients treated with HFNC were treated with an Optiflow device (Fisher&Paykel). Various Bilevel positive airway pressure (BiPAP) devices were used during the study period.

All ventilatory parameters were set according to the treating physicians' preferences.

ELIGIBILITY:
Inclusion Criteria:

* All patients treated with respiratory failure not responding to conventional supplemental oxygen therapy
* Blood venous gas showing partial pressure of carbon dioxide>50 mmHg before beginning therapy with either NIV or HFNC

Exclusion Criteria:

* Lack of records of the primary outcome
* End-of-life care
* Lack of gas before the beginning of NIV or HFNC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated for respiratory II failure in the hospital, including patients treated on the general medical floors, in the emergency department, and in the intensive-care unit.
Sampling Method: Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Failure of initial treatment (combined outcome) | 48 hours post intervention
  Combined outcome of death or intubation or transition to another treatment modality or unplanned resumption of respiratory support
Death at 48h | 48 hours post intervention
  Mortality in the 48h following the initial intervention

SECONDARY OUTCOMES:
Mortality at 7d | 7 days post intervention
  Incidence of death in the 7 days after intervention
Incidence of endotracheal intubation | For the whole length of hospital stay, up to a maximum of one year.
  The incidence of intubation
Length of stay | For the whole length of hospital stay, up to a maximum of one year.
  Duration of stay in the hospital, in days
Duration of endotracheal intubation | For the whole length of hospital stay, up to a maximum of one year.
  Duration (in hours) of the first episode of endotracheal intubation, immediately following the failed intervention
Incidence of intervention change | For the whole length of hospital stay, up to a maximum of one year.
  The incidence of patients who switch from Non-Invasive Ventilation to High-Flow Oxygen, and vice versa, due to treatment failure

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Pavlov, MD, Principal Investigator — Ivan Pavlov MD CP inc
Locations (1):
- Hôpital de Verdun, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No